CLINICAL TRIAL: NCT06148298
Title: Cell-free Chromatin Immunoprecipitation (CfChIP) from Blood Plasma As a Diagnostic and Prognostic Tool in Pancreatic Ductal Adenocarcinoma
Brief Title: Cell-Free DNA Chromatin Immunoprecipitation (ChIP) for Diagnosing Cancer
Status: Recruiting | Type: Observational
Sponsor: University of Central Florida (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00005188
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Cancer of Pancreas
Keywords: cancer; pancreas
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pancreatic Ductal Adenocarcinoma
  Interventions: Other: Non-Human Subject Research study.

INTERVENTIONS:
Other: Non-Human Subject Research study. — This is a Non-Human Subject Research study. There is no intervention. All participants are de-identified.

SUMMARY:
The goal of this research is to use chromatin immunoprecipitation, a method used to study protein-DNA interaction, as a tool to diagnose and prognose pancreatic ductal adenocarcinoma in human samples.

This is a Non-Human Subject Research study. All participants are de-identified.

DETAILED DESCRIPTION:
Pancreatic ductal adenocarcinoma (PDAC) is a neoplastic disease which accounts for "90% of pancreatic malignancies," and has a 5-year survival rate of only 9%. The dismal nature of the PDAC diagnosis, which has a median survival time of about one year, can be attributed in part to late detection. In fact, the Cancer of Pancreas Screening-5 study demonstrated a 73.3% survival rate in participants whose PDAC was found early through surveillance via MRI and endoscopic ultrasound. This eightfold increase in survival rate suggests the inherent efficacy of PDAC screening, however, with the median cost of a full MRI being about $2,000, there is a significant barrier to entry for PDAC screening. As a result, finding a cost-effective alternative to PDAC screening could improve survival rates and lower costs, both directly and indirectly. Liquid biopsy could prove to be a valuable tool in the early diagnosis of PDAC, as it provides a non-invasive way to detect the presence of a disease state such as PDAC. Chromatin immunoprecipitation (ChIP), a type of liquid biopsy used to study protein-DNA interaction, is a promising method at the forefront of cancer research, and has been proven to be capable of detecting tumor-specific transcriptional activity. Additionally, the assay has shown promise in diagnosis and prognosis of disease state. Currently, few (if any) modalities of liquid biopsy in pancreatic cancer use ChIP, and other forms of liquid biopsy have proven to lack sensitivity and specificity. Thus, the aim of this research is to utilize the ChIP assay as a diagnostic and prognostic tool in PDAC by detecting and quantifying tumoral gene expression.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Pancreatic cancer patients

Exclusion Criteria:

* Children may not register
* Persons who are unable to consent may not register

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators want to control for approximate age and have two participants of each gender, and are looking to get 4 without Pancreatic Ductal Adenocarcinoma (PDAC), and 4 of each stage of PDAC (1 through 4).
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Level of c-ERBB1 in blood using Chromatin immunoprecipitation and Reverse transcription-quantitative polymerase chain reaction | 1 year
  Chromatin immunoprecipitation is a method used to study the interaction between DNA and proteins. This makes it a valuable tool for detecting disease state in samples as it allows us to study gene regulation. To put this into practice, DNA is crosslinked to proteins and precipitated out of solution using an antibody. In this case, anti-H3K36me3 was used as it is a marker for active gene regulation which allows for separation of actively transcribed genes. This is synonymous to selecting for a certain disease state that is ongoing. Once this is done, Reverse transcription-quantitative polymerase chain reaction (RT-qPCR) is run on the sample to select for EGFR c-ERBB1, which is an epithelial growth factor (EGFR) mutation which is present in 93% of PDAC cases. Analysis of relative levels of c-ERBB1 should allow for us to diagnose and prognose different stages of PDAC.

CONTACTS AND LOCATIONS:
Overall Officials: Kersten Schroeder, PhD, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No